CLINICAL TRIAL: NCT05447793
Title: Clinical Evalutation of the Effectiveness and Tolerability of Fitostimoline Plus Cream and Gauze vs Connettivina Bio Plus Cream and Gauze in the Treatment of Skin Graft Controlled Randomized Pilot Study
Brief Title: Effectiveness and Tolerability of Fitostimoline Plus vs Connettivina Bio Plus in Skin Graft
Acronym: FP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Barbara Maglione, principal investigator, Federico II University
Other Study IDs: 1808
Record Dates: First submitted 2022-06-30; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Wounds and Injuries; Skin Graft Scar; Skin Graft Complications
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fitostimoline Plus: Formulation in gauzes and cream based on a particular Triticum Vulgare Extract (Rigenase®) and polyhexanide, an antiseptic which does not give any bacterial resistance.
  Interventions: Device: Fitostimoline plus; Device: Connettivina bio plus
- Connettivina Bio Plus: Formulation in gauzes and cream based on hyaluronic acid and silver sulphadiazine.
  Interventions: Device: Fitostimoline plus; Device: Connettivina bio plus

INTERVENTIONS:
Device: Fitostimoline plus — Formulation in gauzes and cream
Device: Connettivina bio plus — Formulation in gauzes and cream

SUMMARY:
Partial thickness skin grafts are widely used to cover large losses of substance secondary to trauma, burns, ulcers, neoplasms.

The donor site (SD), in principle, heals by spontaneous re-epithelialization from the epithelial residues of the skin appendages.

In the post-surgical management of the collection area, in order to optimize treatment, the following are necessary: control of nappy bleeding, management of transudate, avoid superinfection, promote rapid re-epithelialization and pain control.

The objective of the research proposed by us wants to compare two methods of dressing of the SD, one of which involves the use of impregnated gauze and cream with Rigenase and poliesanide (Fitostimoline Plus®) while the other the use of impregnated gauze and cream with hyaluronic acid, sodium salt and 1% silver sulfadiazine (Connettivina Bio Plus®) associated with non-adhesive polyurethane foam (i.e. without adhesive edge, i.e. Mepilex).

The prospective, multicentre study will be conducted at the UOC of Plastic and Reconstructive Surgery of our AOU directed by Prof F. D'Andrea and the UOC of Plastic and Reconstructive Surgery of ASUGI of Trieste directed by Prof Z. Arnez.

To date, there is still no standardized protocol on the wound care of the graft harvesting area. If the literature is evaluated, in fact, large variations in the management of SD are observed with a discrepancy between the practice and the evidence reported in the literature.

The purpose of our research is precisely to review the literature on the effectiveness of dressings at the sampling site level in terms of reducing pain and promoting rapid healing.

DETAILED DESCRIPTION:
The management of the removal site of a partial thickness graft is still a subject of heated debate where, despite the published works, it is still often treated with empirical methods, sometimes which also differ within the same working group. The treatment of AD usually, despite what has been exposed in numerous scientific papers, only involves the use of greasy gauze impregnated with substances that promote re-epithelialization or simple paraffin gauze.

The aim of our research is to compare the effectiveness of bioactive dressings containing Rigenase in association with polyhexanide (PHMB) - Fitostimoline Plus®- with bioactive dressings with hyaluronic acid and Silver sulfadiazine - Connettivina Bio Plus®- in improving the outcome of patients, evaluating:

* cure rate
* the healing times
* the AD infection rate
* pain control / discomfort
* assessment of the scar

RESEARCH OBJECTIVES AND HYPOTHESIS The objective of the study proposed by us is to compare two methods of treating DS; the first involves the use of impregnated gauze and cream containing Rigenase® + polyhexanide; the second is the use of impregnated gauze and sodium salt hyaluronic acid cream. The secondary dressing is a non-adhesive polyurethane foam in both groups.

ELIGIBILITY:
Inclusion Criteria:

* informed consent Age > 18 years

Exclusion Criteria:

* Absence of informed consent Age < 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All pantients aged between 18 and 80 years will be included in the trial if they accept to sign the informed consent.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2022-09-18 (Estimated)

PRIMARY OUTCOMES:
Scarring | one month
  Comparing the two formulations in evaluating the scarring percentage of the lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Maglione, Napoli, Naples, Italy